CLINICAL TRIAL: NCT03480971
Title: A Double Blind, Placebo Controlled Dose Range Finding Study to Assess the Safety, Pharmacokinetics, and Efficacy of Tempol for the Reduction of Severe Mucositis in Head and Neck Cancer Patients Undergoing Combined Radio- and Chemotherapy
Brief Title: Treatment of Radiation and Cisplatin Induced Toxicities with Tempol
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Matrix Biomed, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MBI-04-04
Record Dates: First submitted 2018-03-08; First posted 2018-03-29 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Mucositis; Nephrotoxicity; Ototoxicity
Keywords: cisplatin toxicity
MeSH Terms: conditions — Mucositis; Ototoxicity | interventions — tempol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active 1000 mg Tempol Solution (Active Comparator): Patients will take 1000 mg of Tempol a day for the duration of radiation treatment (6-8 weeks)
  Interventions: Drug: Tempol
- Placebo Solution (Placebo Comparator): Patients will take placebo solution everyday for the duration of radiation treatment (6-8 weeks)
  Interventions: Drug: Placebo Solution

INTERVENTIONS:
Drug: Tempol — Investigational product is Tempol (4-hydroxy-2,2,6,6-tetramethylpiperidine-1-oxyl) oral solution. Tempol solution is an orange-colored, aqueous solution containing 7% Tempol along with xanthan gum, xylitol, aspartame, acesulfame potassium, sodium saccharin, alcohol, peppermint and wintergreen oils.
  Other Names: 4-hydroxy-2,2,6,6-tetramethylpiperidine-1-oxyl
  Arms: Active 1000 mg Tempol Solution
Drug: Placebo Solution — The placebo contains the same excipients as the active product plus FD&C Yellow #6 for color matching.
  Arms: Placebo Solution

SUMMARY:
A 10 week trial to assess the ability of Tempol to prevent and/or reduce toxicities associated with cisplatin and radiation treatment in head and neck cancer patients. Over the course of the 10 week trial, mucositis, nephrotoxicity, and ototoxicity will be monitored and assessed.

DETAILED DESCRIPTION:
One hundred and twenty (120) participants with head and neck cancer are scheduled to undergo combined radio- and chemotherapy (n = 120).

Nearly all (90% to 97%) participants receiving radiotherapy in the head and neck will develop some degree of mucositis. Of these participants treated with radiotherapy with or without chemotherapy, 34% to 43% will present severe mucositis. As a result, the participant's quality of life is affected, hospital admittance rates are higher, the use of total parenteral nutrition is increased and interruption of treatment is more frequent, all of which compromise tumor control. Mucositis causes 9% to 19% of chemotherapy and radiotherapy interruption.

A common chemotherapeutic agent used in head and neck cancer is Cisplatin. Cisplatin (cis- diamminedichloroplatinum(II), CDDP) is an antineoplastic drug used in the treatment of many cancers including testicular cancer, ovarian cancer, bladder cancer, head and neck cancer, esophageal cancer, small and non-small cell lung cancer, breast cancer, cervical cancer, stomach cancer, prostate cancer, brain tumors, neuroblastoma, sarcomas, multiple myeloma, melanoma, mesothelioma, Hodgkin's lymphoma, non-Hodgkin's lymphoma, pancreatic cancer, and thyroid cancer. While toxicities include ototoxicity, gastrotoxicity, myelosuppression, and allergic reactions, the main dose-limiting side effect of cisplatin is nephrotoxicity followed by ototoxicity.

Tempol is a piperidine nitroxide. Nitroxides are a class of stable free radical compounds that protects mammalian cells against numerous toxic agents. Tempol protects normal cells from radiation and cisplatin-induced damage; however, in cancerous or tumor cells, Tempol is reduced to its hydroxylamine form that does not and cannot protect the cells from radiation and cisplatin induced damage. This distinction is of particular importance in the setting of cancer treatment, in which both normal and tumor tissue is exposed to radiation and chemotherapy.

Without using Tempol, both normal cells and cancer cells suffer from toxicity. Tempol is the only known compound to possess this functional duality. This compound has the potential to prevent many of the toxicities associated with cisplatin and radiation treatment including the prevention of mucositis, nephrotoxicity, and ototoxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥18 years of age with medically diagnosed squamous cell cancer of the head and neck (SCCHN);
2. Be scheduled to receive radiotherapy or proton therapy administered with a curative intent;
3. If female and of child bearing potential, be using an effective birth-control method with a history of reliability for the individual participant;
4. If male and of child bearing potential, adequate methods of contraception must be employed including use of condoms with spermicide. No sperm donation for 90 days until after the conclusion of the study;
5. Must be receiving cisplatin for chemotherapy;
6. Be properly informed of the nature and risks of the clinical investigation, comply with all clinical investigation-related procedures, and sign an Informed Consent Form prior to entering the clinical investigation;
7. Must have a score 2 or less on the ECOG performance status;
8. Participant life expectancy ≥ 6 months; and
9. Adequate baseline organ function (hematologic, liver, renal, nutritional and metabolic):

Haematology:

Absolute neutrophil count (ANC) ≥1.5 Hemoglobin ≥ 10 g/dL Platelets ≥ 100,000 per microliter of blood

Hepatic:

Total bilirubin ≤ 2 X (Upper limit normal) ULN Alanine amino transferase (ALT) and Aspartate aminotransferase (AST) ≤5 x ULN

Renal:

Serum creatinine ≤ ULN or, if > ULN calculated creatinine clearance (CrCl) ≥ 60 mL/min.

Nutritional and metabolic:

Urine Albumin < 3.0 mg/dl

Exclusion Criteria:

1. Prior radiotherapy of the head and neck;
2. Have a clinically significant infection defined as any acute viral, bacterial or fungal infection, which requires specific therapy. Anti-infectious therapy must have been completed within 14 days of starting study treatment;
3. Be taking any non-approved therapy for oral mucositis, including β-carotene, tocopherol, laser irradiation, brushing the oral mucosa with silver-nitrate prophylactically, systemic TGF-β (transforming growth factor beta), or systemic KGF (keratinocyte growth factor) during or within 14 days of starting treatment;
4. Be taking mugard;
5. Be taking prostaglandins, pentoxifylline or leucovorin during or within 14 days of starting treatment;
6. Be rinsing with allopurinol, hydrogen peroxide, sucralfate, or chlorhexidine mouthwashes during or within 14 days of starting treatment;
7. Have had a recent, serious, non-malignant medical complication that, in the opinion of the investigator, makes the individual unsuitable for study participation;
8. Have used an investigational drug within 28 days of the initiation of study treatment;
9. Have a history of a positive blood test for HIV;
10. At the time of screening, having a significant active medical illness which, in the opinion of the investigator, would preclude completion of the study;
11. Participants with a treatment plan consisting of chemoradiation followed by further chemotherapy;
12. Participants with body weight less than 35 kg, 77 lbs;
13. Women who are pregnant or who are breastfeeding;
14. Participants with known intolerance to platin drugs;
15. History of insulin-dependent Diabetes Mellitus; and
16. Participants with Hepatitis B/C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-05-13 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Mucositis | 10 weeks
  To determine the efficacy of Tempol in reducing the incidence severe mucositis defined as grade 3 or 4 on the World Health Organization (WHO) scale.
  The incidence will measure the number of patients who experience grade 3 or 4 mucositis according to the World Health Organization (WHO) scale. A reduction in the number of patients who receive grade 3 or 4 mucositis over the course of the treatment is considered a positive change in incidence.

SECONDARY OUTCOMES:
Mucositis | 10 weeks
  To determine the efficacy of Tempol in reducing the duration severe mucositis defined as grade 3 or 4 on the World Health Organization (WHO) scale.
  This duration will be measured by total number of days number a patient experiences grade 3 or 4 mucositis according to the World Health Organization (WHO) scale. A reduction in the total number of days a patient receives grade 3 or 4 mucositis over the course of the treatment is considered a positive change in duration.
Nephrotoxicity | 10 weeks
  Reduction in Serum Creatinine levels in active arm versus placebo arm.
Nephrotoxicity | 10 weeks
  Reduction in Blood Urea Nitrogen levels in active arm versus placebo arm.
Mucositis | 10 weeks
  To determine the efficacy of Tempol in reducing the time to onset of grades 1-4 mucositis on the World Health Organization (WHO) scale.
  This time to onset will measure the number of days after exposure to cisplatin before a patient experiences grade 1 through 4 mucositis according to the World Health Organization (WHO) scale. An increase in the total number of days before a patient receives grade 1 through 4 mucositis after cisplatin exposure is considered a positive change in time to onset.

CONTACTS AND LOCATIONS:
Overall Officials: Benji Crane, Study Director — Matrix Biomed, Inc.
Locations (9):
- United States (9):
  - UCSD, La Jolla, California
  - Mercy Medical Center, Merced, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Central Coast Medical Oncology, Santa Maria, California
  - Mission Hope Health Center, Santa Maria, California
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arany I, Safirstein RL. Cisplatin nephrotoxicity. Semin Nephrol. 2003 Sep;23(5):460-4. doi: 10.1016/s0270-9295(03)00089-5. PMID 13680535
- [Background] Ahmed LA, Shehata NI, Abdelkader NF, Khattab MM. Tempol, a superoxide dismutase mimetic agent, ameliorates cisplatin-induced nephrotoxicity through alleviation of mitochondrial dysfunction in mice. PLoS One. 2014 Oct 1;9(10):e108889. doi: 10.1371/journal.pone.0108889. eCollection 2014. PMID 25271439
- [Background] Scully C, Sonis S, Diz PD. Oral mucositis. Oral Dis. 2006 May;12(3):229-41. doi: 10.1111/j.1601-0825.2006.01258.x. PMID 16700732
- [Background] Hartmann JT, Lipp HP. Toxicity of platinum compounds. Expert Opin Pharmacother. 2003 Jun;4(6):889-901. doi: 10.1517/14656566.4.6.889. PMID 12783586
- [Background] Sastry J, Kellie SJ. Severe neurotoxicity, ototoxicity and nephrotoxicity following high-dose cisplatin and amifostine. Pediatr Hematol Oncol. 2005 Jul-Aug;22(5):441-5. doi: 10.1080/08880010590964381. PMID 16020136
- [Background] Samuni A, Winkelsberg D, Pinson A, Hahn SM, Mitchell JB, Russo A. Nitroxide stable radicals protect beating cardiomyocytes against oxidative damage. J Clin Invest. 1991 May;87(5):1526-30. doi: 10.1172/JCI115163. PMID 1850756
- [Background] Samuni A, Mitchell JB, DeGraff W, Krishna CM, Samuni U, Russo A. Nitroxide SOD-mimics: modes of action. Free Radic Res Commun. 1991;12-13 Pt 1:187-94. doi: 10.3109/10715769109145785. PMID 1649088
- [Background] Samuni A, Krishna CM, Mitchell JB, Collins CR, Russo A. Superoxide reaction with nitroxides. Free Radic Res Commun. 1990;9(3-6):241-9. doi: 10.3109/10715769009145682. PMID 2167262
- [Background] Mitchell JB, Anver MR, Sowers AL, Rosenberg PS, Figueroa M, Thetford A, Krishna MC, Albert PS, Cook JA. The antioxidant tempol reduces carcinogenesis and enhances survival in mice when administered after nonlethal total body radiation. Cancer Res. 2012 Sep 15;72(18):4846-55. doi: 10.1158/0008-5472.CAN-12-1879. Epub 2012 Jul 17. PMID 22805306